CLINICAL TRIAL: NCT04220229
Title: A Phase 1/2 Study of Neoadjuvant Cabozantinib in Combination With Radiation Therapy for Sarcomas of the Extremities
Brief Title: Cabozantinib With Radiation Therapy for the Treatment of Sarcomas of the Extremities
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Terminated due to end of funding
Sponsor: University of Washington (Other)
Collaborators: Exelixis (Industry)
Responsible Party: Principal Investigator, Lee Duncan Cranmer, Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1003562; NCI-2019-08661 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10051 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2020-01-03; First posted 2020-01-07 (Actual); Results first posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-06

CONDITIONS: Sarcoma of the Extremity; Stage I Soft Tissue Sarcoma of the Trunk and Extremities; Stage IA Soft Tissue Sarcoma of the Trunk and Extremities; Stage IB Soft Tissue Sarcoma of the Trunk and Extremities; Stage II Soft Tissue Sarcoma of the Trunk and Extremities
Keywords: Soft Tissue
MeSH Terms: interventions — cabozantinib; Succinic Acid; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (cabozantinib S-malate, radiation therapy) (Experimental): Patients receive cabozantinib S-malate PO QD on days 1-21. Cycles repeat every 21 days until the completion of radiation therapy in the absence of disease progression or unacceptable toxicity. Beginning cycle 1 day 8, patients also undergo standard of care radiation therapy for 5-6 weeks.
  Interventions: Drug: Cabozantinib S-malate; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Cabozantinib S-malate — Given PO
  Other Names: 1140909-48-3; BMS-907351; Butanedioic acid; Cabometyx; Cometriq
Radiation: Radiation Therapy — Undergo standard of care radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; irradiated; Irradiation; RADIATION; NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation

SUMMARY:
This phase I/II trial studies the side effects and best dose of cabozantinib when given with radiation therapy and how well it works in treating patients with sarcoma of the extremities. Cabozantinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving cabozantinib with radiation therapy may make the tumors smaller and reduce the amount of normal tissue that needs to be removed.

DETAILED DESCRIPTION:
OUTLINE: This is a phase I, dose-escalation study of cabozantinib followed by a phase II, dose-expansion study.

Patients receive cabozantinib S-malate orally (PO) once daily (QD) on days 1-21. Cycles repeat every 21 days until the completion of radiation therapy in the absence of disease progression or unacceptable toxicity. Beginning Cycle 1 Day 8, patients also undergo standard of care radiation therapy for 5-6 weeks.

After completion of study treatment, patients are followed up at 30 days, every 12 weeks for up to 1 year, then every 6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects, >= 18 years old, must have a histologically confirmed diagnosis of sarcomas of the extremities (which may include gluteal muscle involvement) for which neoadjuvant radiation therapy followed by surgical resection is a planned intervention

  * Subjects whose bowel cannot be completely protected from radiation exposure due to primary tumor location (e.g., proximal lower extremity) will be excluded
* Subjects must have one or more measurable target lesions by RECIST version (v) 1.1, assessed via computed tomography (CT) scan or magnetic resonance imaging (MRI)
* At the time of study enrollment, subjects must have a tumor burden that is judged to be surgically resectable
* Absolute neutrophil count (ANC) >= 1500/mm^3 (>= 1.5 GI/L) without granulocyte colony-stimulating factor support in the last 28 days
* White blood cell count >= 2500/mm^3 (>= 2.5 GI/L)
* Platelets >= 100,000/mm^3 (>=100 GI/L) without transfusion in the last 28 days
* Hemoglobin >= 9 g/dL (>= 90 g/L) without transfusion in the last 28 days
* Alanine aminotransferase (ALT), aspartate aminotransferase (AST) =< 3 X upper limit of normal (ULN)
* Alkaline phosphatase (ALP) =< 3 X upper limit of normal (ULN)

  * ALP =< 5 X ULN is permitted in subjects with documented bone metastases (phase 1 only)
* Total bilirubin =< 1.5 x ULN (for subjects with Gilbert's disease =< 3 X ULN)
* Serum albumin >= 2.8 g/dl
* Serum creatinine =< 2.0 x ULN or calculated creatinine clearance >= 30 mL/min (>= 0.5 mL/sec) using the Cockcroft-Gault equation
* Urine protein/creatinine ratio (UPCR) =< 1 mg/mg (=< 113.2 mg/mmol)
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Male or non-pregnant and non-breast feeding female:

  * Females of child-bearing potential must agree to use highly effective contraception without interruption from initiation of therapy and while on study medication and have a negative serum pregnancy test (beta-human chorionic gonadotropin [B-hCG]) result at screening and agree to ongoing pregnancy testing during the study, and at the end of study treatment. A highly effective method of contraception is defined as one that results in a low failure rate (that is, < 1% per year), when used consistently and correctly, such as implants, injectables, combined oral contraceptives, some intrauterine contraceptive devices, sexual abstinence, or a vasectomized partner
  * Male subjects must practice abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study
* Life expectancy of > 3 months, as determined by the investigator
* Ability to understand and sign informed consent
* Willingness and ability to comply with scheduled visits, laboratory tests, and other study procedures

Exclusion Criteria:

* Receipt of any type of cytotoxic, biologic or other systemic anticancer therapy (including investigational) for the investigational diagnosis
* Receipt of any prior radiation therapy for the investigational diagnosis
* Known central nervous system (CNS) metastases
* Concomitant anticoagulation with oral anticoagulants(e.g., warfarin, direct thrombin and factor Xa inhibitors) or platelet inhibitors (e.g., clopidogrel). Allowed anticoagulants are the following:

  * Low-dose aspirin for cardioprotection (per local applicable guidelines) is permitted
  * Low-dose low molecular weight heparins (LMWH) are permitted
  * Anticoagulation with therapeutic doses of LMWH is allowed in subjects without known brain metastases who are on a stable dose of LMWH for at least 6 weeks before first dose of study treatment, and who have had no clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor. Subjects with hemoptysis, central nervous system hemorrhage or gastrointestinal hemorrhage within the last 6 months prior to treatment are excluded
* The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  * Cardiovascular disorders:

    * Congestive heart failure New York Heart Association Class 3 or 4, unstable angina pectoris, serious cardiac arrhythmias
    * Uncontrolled hypertension defined as sustained blood pressure (BP) > 150 mm Hg systolic or > 100 mm Hg diastolic despite optimal anti-hypertensive treatment
    * Stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic event, or thromboembolic event (e.g., deep venous thrombosis, pulmonary embolism) within 6 months before first dose.
  * Uncontrolled serious medical or psychiatric illness
  * Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation:

    * The subject has evidence of tumor invading the GI tract, active peptic ulcer disease, inflammatory bowel disease (e.g., Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis, acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction
    * Abdominal fistula, GI perforation, bowel obstruction, or intra-abdominal abscess within 6 months before first dose
    * Note: Complete healing of an intra-abdominal abscess must be confirmed before first dose
  * Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (e.g., pulmonary hemorrhage) within 12 weeks before first dose
  * Cavitating pulmonary lesion(s) or known endotracheal or endobronchial disease manifestation
  * Lesions invading or encasing any major blood vessels
  * Other clinically significant disorders that would preclude safe study participation

    * Serious non-healing wound/ulcer/bone fracture
    * Uncompensated/symptomatic hypothyroidism
    * Moderate to severe hepatic impairment (Child-Pugh B or C)
* Major surgery (e.g., GI surgery, removal or biopsy of brain metastasis) within 8 weeks before first dose of study treatment. Complete wound healing from major surgery must have occurred at least 30 days before first dose, and from minor surgery (e.g., simple excision, tooth extraction) at least 10 days before first dose. Subjects with clinically relevant ongoing complications from prior surgery are not eligible
* Corrected QT interval calculated by the Bazett's formula (corrected QT [QTc]) > 480 ms per electrocardiogram (ECG) within 28 days before first dose of study treatment

  * Note: If a single ECG shows a QTc with an absolute value > 480 ms, two additional ECGs at intervals of approximately 3 min must be performed within 30 min after the initial ECG, and the average of these three consecutive results for QTc will be used to determine eligibility
* Pregnant or lactating females
* Inability to swallow tablets
* Previously identified allergy or hypersensitivity to components of the study treatment formulations
* Diagnosis of another malignancy within 2 years before first dose of study treatment, except for superficial skin cancers, or localized, low-grade tumors deemed cured and not treated with systemic therapy
* Concurrent use of medications (especially those interacting with CYP3A417) that potentially interact unsafely with cabozantinib which cannot be discontinued or substituted
* Subjects with a sarcoma which has other, defined treatments or biology distinctly different from those of soft tissue sarcomas in general. Including, but not limited to, Ewing's sarcoma, rhabdomyosarcoma, gastrointestinal stromal tumors, Kaposi's sarcoma, Wilms' tumor
* Transfusion of blood product or granulocyte-colony stimulating factor (G-CSF) support factor within the last 28 days
* Recent infection requiring systemic anti-infective treatment that was completed =< 14 days prior to enrollment (except for uncomplicated urinary tract infection or upper respiratory tract infection)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee Cranmer, MD, PhD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vatner R, James CD, Sathiaseelan V, Bondra KM, Kalapurakal JA, Houghton PJ. Radiation therapy and molecular-targeted agents in preclinical testing for immunotherapy, brain tumors, and sarcomas: Opportunities and challenges. Pediatr Blood Cancer. 2021 May;68 Suppl 2:e28439. doi: 10.1002/pbc.28439. Epub 2020 Aug 22. PMID 32827353

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study was terminated prior to enrolling participants in Phase II portion of study.
Groups:
- Treatment (40 mg Cabozantinib S-malate, Radiation Therapy): Patients receive 40 mg cabozantinib S-malate PO QD on days 1-21. Cycles repeat every 21 days until the completion of radiation therapy in the absence of disease progression or unacceptable toxicity. Beginning cycle 1 day 8, patients also undergo standard of care radiation therapy for 5-6 weeks.
  Cabozantinib S-malate: Given PO
  Radiation Therapy: Undergo standard of care radiation therapy
- Treatment (60 mg Cabozantinib S-malate, Radiation Therapy): Patients receive 60 mg cabozantinib S-malate PO QD on days 1-21. Cycles repeat every 21 days until the completion of radiation therapy in the absence of disease progression or unacceptable toxicity. Beginning cycle 1 day 8, patients also undergo standard of care radiation therapy for 5-6 weeks.
  Cabozantinib S-malate: Given PO
  Radiation Therapy: Undergo standard of care radiation therapy
Period: Overall Study
Arm/Group | Treatment (40 mg Cabozantinib S-malate, Radiation Therapy) | Treatment (60 mg Cabozantinib S-malate, Radiation Therapy)
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 1: 40 mg Cabozantinib S-malate, Radiation Therapy: Patients receive 40 mg cabozantinib S-malate PO QD on days 1-21. Cycles repeat every 21 days until the completion of radiation therapy in the absence of disease progression or unacceptable toxicity. Beginning cycle 1 day 8, patients also undergo standard of care radiation therapy for 5-6 weeks.
  Cabozantinib S-malate: Given PO
  Radiation Therapy: Undergo standard of care radiation therapy
- Phase 1: 60 mg Cabozantinib S-malate, Radiation Therapy: Patients receive 60 mg cabozantinib S-malate PO QD on days 1-21. Cycles repeat every 21 days until the completion of radiation therapy in the absence of disease progression or unacceptable toxicity. Beginning cycle 1 day 8, patients also undergo standard of care radiation therapy for 5-6 weeks.
  Cabozantinib S-malate: Given PO
  Radiation Therapy: Undergo standard of care radiation therapy
- Total: Total of all reporting groups
Arm/Group | Phase 1: 40 mg Cabozantinib S-malate, Radiation Therapy | Phase 1: 60 mg Cabozantinib S-malate, Radiation Therapy | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Customized [Count of Participants; unit: Participants]
  18-29 | 0 | 0 | 0
  30-39 | 0 | 0 | 0
  40-49 | 1 | 1 | 2
  50-59 | 2 | 1 | 3
  60-69 | 0 | 1 | 1
  70+ | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase 2 Dose of Cabozantinib S-malate (Cabozantinib) (Phase I)
Description: Cabozantinib treatment begins 8 days prior to initiation of radiation therapy and continues through completion of radiation therapy.
Time Frame: Up to 21 days
Measure: Number; unit: mg
Arm/Group | Treatment (Cabozantinib S-malate, Radiation Therapy)
Number analyzed (Participants) | 6
mg | 60

2. Primary Outcome: Rate of Relapse (Phase II)
Description: No patients were enrolled in Phase II portion of study - outcome measure based on Phase I patients.
Time Frame: At 12 months after treatment initiation
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1: 40 mg Cabozantinib S-malate, Radiation Therapy | Phase 1: 60 mg Cabozantinib S-malate, Radiation Therapy
Number analyzed (Participants) | 3 | 3
percentage of participants | 0 [0 to 71] | 33 [0 to 91]

3. Secondary Outcome: Rate of Pathologic Response(>90%)
Description: Evaluated utilizing the Exact Clopper-Pearson method.
Time Frame: Up to 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1: 40 mg Cabozantinib S-malate, Radiation Therapy | Phase 1: 60 mg Cabozantinib S-malate, Radiation Therapy
Number analyzed (Participants) | 3 | 3
percentage of participants | 0 [0 to 71] | 33 [0 to 91]

4. Secondary Outcome: Rate of Surgical Excision With Negative Margins
Description: Evaluated utilizing the Exact Clopper-Pearson method.
Time Frame: Up to 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Phase 1: 60 mg Cabozantinib S-malate, Radiation Therapy: Patients receive 60 cabozantinib S-malate PO QD on days 1-21. Cycles repeat every 21 days until the completion of radiation therapy in the absence of disease progression or unacceptable toxicity. Beginning cycle 1 day 8, patients also undergo standard of care radiation therapy for 5-6 weeks.
  Cabozantinib S-malate: Given PO
  Radiation Therapy: Undergo standard of care radiation therapy
Arm/Group | Phase 1: 40 mg Cabozantinib S-malate, Radiation Therapy | Phase 1: 60 mg Cabozantinib S-malate, Radiation Therapy
Number analyzed (Participants) | 3 | 3
percentage of participants | 100 [29 to 100] | 100 [29 to 100]

5. Secondary Outcome: Objective Response Rate
Description: Will be defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria. Includes those who had complete response and partial response.
Time Frame: Up to 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Phase 1: 60 mg Cabozantinib S-malate, Radiation Therapy: Patients receive cabozantinib S-malate PO QD on days 1-21. Cycles repeat every 21 days until the completion of radiation therapy in the absence of disease progression or unacceptable toxicity. Beginning cycle 1 day 8, patients also undergo standard of care radiation therapy for 5-6 weeks.
  Cabozantinib S-malate: Given PO
  Radiation Therapy: Undergo standard of care radiation therapy
Arm/Group | Phase 1: 40 mg Cabozantinib S-malate, Radiation Therapy | Phase 1: 60 mg Cabozantinib S-malate, Radiation Therapy
Number analyzed (Participants) | 3 | 3
percentage of participants | 0 [0 to 71] | 0 [0 to 71]

6. Secondary Outcome: Rate of Local Relapse
Description: Evaluated utilizing the Exact Clopper-Pearson method.
Time Frame: Up to 3 years
Measure: Number (95% Confidence Interval); unit: precentage of participants
Arm/Group | Phase 1: 40 mg Cabozantinib S-malate, Radiation Therapy | Phase 1: 60 mg Cabozantinib S-malate, Radiation Therapy
Number analyzed (Participants) | 3 | 3
precentage of participants | 0 [0 to 71] | 0 [0 to 71]

7. Secondary Outcome: Rate of Distant Relapse
Description: Evaluated utilizing the Exact Clopper-Pearson method.
Time Frame: Up to 3 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1: 40 mg Cabozantinib S-malate, Radiation Therapy | Phase 1: 60 mg Cabozantinib S-malate, Radiation Therapy
Number analyzed (Participants) | 3 | 3
percentage of participants | 0 [0 to 71] | 66 [9 to 99]

8. Secondary Outcome: Relapse-free Survival
Description: Evaluated utilizing the Exact Clopper-Pearson method.
Time Frame: Up to 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1: 40 mg Cabozantinib S-malate, Radiation Therapy | Phase 1: 60 mg Cabozantinib S-malate, Radiation Therapy
Number analyzed (Participants) | 3 | 3
percentage of participants | 100 [29 to 100] | 66 [9 to 99]

9. Secondary Outcome: Overall Survival
Description: Evaluated utilizing the Exact Clopper-Pearson method.
Time Frame: Up to 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1: 40 mg Cabozantinib S-malate, Radiation Therapy | Phase 1: 60 mg Cabozantinib S-malate, Radiation Therapy
Number analyzed (Participants) | 3 | 3
percentage of participants | 100 [29 to 100] | 100 [29 to 100]

10. Secondary Outcome: Incidence of Adverse Events - Treatment-related Adverse Events (AEs) Experienced by Participants Evaluated by CTCAE 5.0 and Determined to be Possibly Related, Probably Related, or Definitely Related to Cabozantinib.
Description: Adverse events will be graded by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0.
Time Frame: Up to 30 days after last dose of investigational product (an average of up to 12 weeks)
Measure: Number; unit: adverse events experienced
Arm/Group | Phase 1: 40 mg Cabozantinib S-malate, Radiation Therapy | Phase 1: 60 mg Cabozantinib S-malate, Radiation Therapy
Number analyzed (Participants) | 3 | 3
adverse events experienced
  Grade 1 | 20 | 24
  Grade 2 | 7 | 5
  Grade 3 | 2 | 3
  Grade 4 | 0 | 0
  Grade 5 | 0 | 0

11. Secondary Outcome: Rate of Treatment Discontinuation Prior to Neoadjuvant Radiation Therapy
Description: Evaluated utilizing the Exact Clopper-Pearson method.
Time Frame: Up to 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1: 40 mg Cabozantinib S-malate, Radiation Therapy | Phase 1: 60 mg Cabozantinib S-malate, Radiation Therapy
Number analyzed (Participants) | 3 | 3
percentage of participants | 0 [0 to 71] | 0 [0 to 71]

ADVERSE EVENTS:
Time Frame: Adverse events will be collected up to 30 days post last dose of study treatment, for an average of up to 12 weeks. All-cause mortality was assessed until study end, for an average of 112 weeks.
Arm/Group | Phase 1: 40 mg Cabozantinib S-malate, Radiation Therapy | Phase 1: 60 mg Cabozantinib S-malate, Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 1/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: 40 mg Cabozantinib S-malate, Radiation Therapy (N=3) | Phase 1: 60 mg Cabozantinib S-malate, Radiation Therapy (N=3)
Mucositis oral (Gastrointestinal disorders) | 3 (3) | 3 (3)
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Anosmia (Nervous system disorders) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (3) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Edema face (General disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (4) | 3 (3)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other (General disorders) | 1 (1) | 0 (0)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hair color changes (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperlipidemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertension (Surgical and medical procedures) | 2 (3) | 3 (4)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Muscle Cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nervous system disorders - Other (Nervous system disorders) | 0 (0) | 1 (1)
Neutrophil count decreased (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Papulopustular rash (Infections and infestations) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Periorbital edema (Eye disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (General disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Psychiatric disorders - Other (Psychiatric disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Weight loss (Investigations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-04): https://cdn.clinicaltrials.gov/large-docs/29/NCT04220229/Prot_SAP_001.pdf
  • Informed Consent Form (2023-03-09): https://cdn.clinicaltrials.gov/large-docs/29/NCT04220229/ICF_000.pdf